CLINICAL TRIAL: NCT07012603
Title: External Oblique and Rectus Abdominis Plane (EXORA) Block for Postoperative Analgesia in Patients Undergoing Umbilical Hernia Repair: A Randomized Controlled Trial
Brief Title: External Oblique and Rectus Abdominis Plane (EXORA) Block for Postoperative Analgesia in Patients Undergoing Umbilical Hernia Repair
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Mohammed Said ElSharkawy, Lecturer of Anesthesiology, Surgical Intensive Care and Pain Medicine, Faculty of Medicine, Tanta University, Tanta, Egypt., Tanta University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 36264PR1207/5/25
Record Dates: First submitted 2025-05-31; First posted 2025-06-10 (Actual); Last update posted 2025-06-11 (Actual); Status verified 2025-06

CONDITIONS: External Oblique and Rectus Abdominis Plane; Postoperative Analgesia; Umbilical Hernia Repair
MeSH Terms: interventions — Dental Occlusion

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- EXORA block group (Experimental): Patients will receive an external oblique and rectus abdominis plane (EXORA) block using 20 mL of bupivacaine 0.25%.
  Interventions: Other: External oblique and rectus abdominis plane (EXORA) block
- Control group (Sham Comparator): Patients will receive a sham block using 20 mL of normal saline as a control group.
  Interventions: Other: Sham block

INTERVENTIONS:
Other: External oblique and rectus abdominis plane (EXORA) block — Patients will receive an external oblique and rectus abdominis plane (EXORA) block using 20 mL of bupivacaine 0.25%.
  Arms: EXORA block group
Other: Sham block — Patients will receive a sham block using 20 mL of normal saline as a control group.
  Arms: Control group

SUMMARY:
This study aims to evaluate the effect of the external oblique and rectus abdominis plane (EXORA) block for postoperative analgesia in patients undergoing umbilical hernia repair.

DETAILED DESCRIPTION:
Umbilical hernias account for approximately 6-14% of adult abdominal wall hernias. These hernias are typically acquired and are mainly caused by increased abdominal pressure. Umbilical hernias do not heal on their own and usually require surgical intervention.

The external oblique and rectus abdominis plane (EXORA) block is an emerging technique providing a sensory block to the anterolateral abdominal wall. The EXORA block involves local anaesthetic injection into the fascial plane between the external oblique and rectus abdominis muscles. This method provides better dermatomal coverage, making the EXORA block particularly effective in the treatment of somatic pain in the anterolateral area of the upper and middle abdomen.

ELIGIBILITY:
Inclusion Criteria:

* Age from 18 to 65 years.
* Both sexes.
* American Society of Anesthesiology (ASA) physical status I-II.
* Undergoing umbilical hernia repair.

Exclusion Criteria:

* History of allergies to local anesthetics.
* Bleeding or coagulation disorders.
* Anatomical abnormalities.
* Psychiatric and neurological disorders.
* Local infection at the site of injection.
* Complicated hernial defects [strangulated, incarcerated, or obstructed cases].

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-06-10 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Total morphine consumption | 24 hours postoperatively
  Rescue analgesia of morphine will be given as 5 mg bolus if the numeric rating scale (NRS) > 3 to be repeated after 30 min if pain persists until the NRS < 4.

SECONDARY OUTCOMES:
Time to the 1st rescue analgesia | 24 hours postoperatively
  Time to the first request for the rescue analgesia (time from the end of surgery to first dose of morphine administrated).
Intraoperative fentanyl consumption | Intraoperatively
  Additional fentanyl bolus dosages of 1 µg/kg IV will be administered if heart rate or mean arterial blood pressure elevated more than 20% of the baseline (after exclusion of other causes than pain).
Degree of pain | 24 hours postoperatively
  Each patient will be instructed about postoperative pain assessment with the numeric rating scale (NRS) score. NRS (0 represents "no pain" while 10 represents "the worst pain imaginable"). NRS will be assessed at post-anesthesia care unit (PACU), 2, 4, 6, 8, 12, and 24 h postoperatively.
Mean arterial pressure | Till the end of surgery (Up to 2 hours)
  Mean arterial pressure will be recorded preoperatively and every 30 minutes till the end of surgery.
Heart rate | Till the end of surgery (Up to 2 hours)
  Heart rate will be recorded preoperatively and every 30 minutes till the end of surgery.
Incidence of adverse events | 24 hours postoperatively
  Incidence of adverse events such as bradycardia, hypotension, nausea, vomiting, respiratory depression, or any other complication will be recorded.

CONTACTS AND LOCATIONS:
Locations (1):
- Tanta University, Tanta, El-Gharbia, Egypt

IPD SHARING:
Plan to Share IPD: Yes
The data will be available upon a reasonable request from the corresponding author after the end of study for one year.
Supporting Information: Study Protocol
Time Frame: After the end of study for one year.
Access Criteria: The data will be available upon a reasonable request from the corresponding author.